CLINICAL TRIAL: NCT03454737
Title: Treatment of Refractory Patellar Tendinopathy With Mesenquimal Trunk Cells. Comparative Study With PRP.
Acronym: TENDO
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Institut de Terapia Regenerativa Tissular (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MSC-TENDO-2015; 2016-001262-28 (EudraCT Number)
Record Dates: First submitted 2018-01-04; First posted 2018-03-06 (Actual); Last update posted 2018-12-19 (Actual); Status verified 2018-03

CONDITIONS: Patellar Tendinopathy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- mesenchymal stem cells (Experimental)
  Interventions: Procedure: mesenchymal stem cells
- Pure platelet-rich plasma (Active Comparator)
  Interventions: Procedure: Pure platelet-rich plasma

INTERVENTIONS:
Procedure: mesenchymal stem cells — Autologous bone marrow aspiration is used as a cellular source to obtain MSVs and is subjected to the protocolized anticoagulant procedure. After checking the perfect condition of the shipment and the correct completion of the documentation that accompanies it, the processing of the bone marrow will be carried out.
  The processing of the bone marrow will be done in the Cell Therapy Unit of the IBGM under NCF, within 24 hours of the completion of the aspiration
  Arms: mesenchymal stem cells
Procedure: Pure platelet-rich plasma — Under aseptic conditions, in surgical medium, 6 ml of P-PRP will be obtained from 36 ml of autologous peripheral venous blood sample.
  The plasma coagulation will be activated by the addition of Cl2Ca at a concentration of 5%.
  Arms: Pure platelet-rich plasma

SUMMARY:
This is a clinical trial, unicentric, prospective, controlled, randomized, double blind during the experimental phase A.

In the experimental phase B, it is contemplated to administer the experimental treatment to the subjects included in the group treated with P-PRP in the event that the first treatment would be significantly more effective, both from a clinical and regenerative point of view

DETAILED DESCRIPTION:
* Main objective

  1. Confirm the presence of patellar tendon gap regeneration after the peritendinous and intratendinous infusion of MSV and compare it with the P-PRP group, evaluated by ECO, NMR and UTC.
  2. To evaluate the clinical efficacy of infusion of MSC in refractory patellar tendinopathy compared with the P-PRP group through the subjective clinical evolution of the patient, the EVA and VISA-P questionnaires and the strength of the extensor muscle group measured by dynamometry.
* Secondary objective 1. To evaluate the feasibility and safety of the advanced therapy medication MSV and P-PRP when applied by percutaneous infusion into the body of the patellar tendinosis, verifying that each of the procedures established in the protocol is feasible and recording the possible adverse effects related with both treatments and adverse events arising during the period of the clinical trial, whether or not related to it

ELIGIBILITY:
Inclusion Criteria:

1. Male sex with ages between 18 and 48 years.
2. Pain in the patellar tendon, located in the patellar insertion area, of more than 4 months of duration that does not show significant improvement after conservative treatments such as rest, analgesia, physiotherapy and / or infiltration.
3. Ultrasound image that confirms, both static and dynamic, the loss of the fibrillar structure of the proximal part of the patellar tendon, its thickening and a hypoechoic lesion compatible with gap ≥3mm.
4. MRI of the patellar tendon in T2 FAT SAT sequence (fat saturation) that shows a gap ≥3mm in longitudinal diameter in the proximal insertion.
5. Informed Consent in writing and signed by the patient.
6. The patient is able to understand the nature of the study.

Exclusion Criteria:

1. Patient under 18 years of age (or legally dependent) and over 48 years of age.
2. MRI with grade III-IV intra-articular pathology of all compartments of the knee and / or cruciate ligament injury
3. Local treatment with corticosteroids during the last year
4. Local treatment with PRP during the last 6 months.
5. Present infection (no local or systemic infectious signs should be evidenced).
6. Patients presenting positive serology in front of:

   HIV 1 and 2, Hepatitis B (HBsAg, HBcAc), Hepatitis C (Anti-HCV-Ab), Lúes.
7. Congenital or evolutive diseases that translate malformation and / or significant deformations of the knee and condition difficulties of application and evaluation of the results.
8. Weight overload expressed in body mass index (BMI) greater than 30.5 (obesity grade II). Being BMI = mass (Kg): (height (m)) 2
9. Active neoplastic disease.
10. Active immunosuppressive states.
11. Simultaneous participation in another clinical trial or treatment with another product in the Research phase in the 30 days prior to inclusion in the study.
12. Other pathologies or circumstances that compromise participation in the study according to medical criteri

Ages: 18 Years to 48 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2017-12-13 (Actual); Primary Completion 2019-06-20 (Estimated); Study Completion 2020-12-14 (Estimated)

PRIMARY OUTCOMES:
Improvement in the tendon ecotexture | 24 months
  The patellar tendon will be examined longitudinally and transversely using gray scale and color, exerting a minimum pressure with the probe. Images will be recorded in static and dynamic formats to develop a consensus of the findings.

SECONDARY OUTCOMES:
Presence of patellar tendon regeneration by the peritendinous and intratendinous infusion of MSV patellar tendinopathy compared to the P-PRP group | 24 months
  Using ECO, RMN and UTC (Ultrasound Tissue Characterisation)
the strength of the extensor muscle group | 24 months
  using dynamometry.
subjective clinical evolution of the patient | 24 months
  Using EVA and VISA-P (Victorian Institute of Sport Assessment (patelar)) questionnaries.
strength of the extensor muscle group | 24 months
  Using dynamometry

CONTACTS AND LOCATIONS:
Overall Officials: Gil Rodas, MD, Principal Investigator — Centro Médico Teknon
Locations (1):
- Institut de Terapia Regenerativa Tissular, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Rodas G, Soler-Rich R, Rius-Tarruella J, Alomar X, Balius R, Orozco L, Masci L, Maffulli N. Effect of Autologous Expanded Bone Marrow Mesenchymal Stem Cells or Leukocyte-Poor Platelet-Rich Plasma in Chronic Patellar Tendinopathy (With Gap >3 mm): Preliminary Outcomes After 6 Months of a Double-Blind, Randomized, Prospective Study. Am J Sports Med. 2021 May;49(6):1492-1504. doi: 10.1177/0363546521998725. Epub 2021 Mar 30. PMID 33783227
- [Derived] Rodas G, Soler R, Balius R, Alomar X, Peirau X, Alberca M, Sanchez A, Sancho JG, Rodellar C, Romero A, Masci L, Orozco L, Maffulli N. Autologous bone marrow expanded mesenchymal stem cells in patellar tendinopathy: protocol for a phase I/II, single-centre, randomized with active control PRP, double-blinded clinical trial. J Orthop Surg Res. 2019 Dec 16;14(1):441. doi: 10.1186/s13018-019-1477-2. PMID 31842921